CLINICAL TRIAL: NCT05928013
Title: Neuropathy Evaluation Using the Vibration Function of a Mobile Phone - the NERVE Study
Brief Title: Neuropathy Evaluation Using the Vibration of a Mobile Phone
Acronym: NERVE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospitals Dorset NHS Foundation Trust (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: NERVE
Record Dates: First submitted 2023-05-25; First posted 2023-07-03 (Actual); Last update posted 2025-02-21 (Actual); Status verified 2025-02

CONDITIONS: Diabetic Foot
MeSH Terms: conditions — Diabetic Foot

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Person With Diabetes (Experimental): A health care professional will conduct the vibration perception threshold testing using both the Neurothesiometer and NERVE diagnostic testing on the person with diabetes. The person with diabetes will conduct the vibration perception threshold testing using the NERVE device. There is an option for a carer/buddy to conduct the vibration perception threshold testing with the NERVE device on the person with diabetes.
  Interventions: Diagnostic Test: Neurothesiometer; Diagnostic Test: NERVE

INTERVENTIONS:
Diagnostic Test: Neurothesiometer — The 'gold standard' device for Vibration Perception Threshold testing
Diagnostic Test: NERVE — The experimental device for Vibration Perception Threshold testing developed by the project team

SUMMARY:
A single centre validation/method comparison study of the experimental NERVE device for the measurement of vibration perception threshold against the established 'Neurothesiometer' device, evaluating agreement and reliability. It will also include collecting feedback from patients, carers and clinicians on the usability of the device

ELIGIBILITY:
Inclusion Criteria:

* Formally Diagnosed With Diabetes

Exclusion Criteria:

* 1. Un- willing or un-able to provide free informed consent (no time limit)
* 2. Un-willing or un-able to comply with all protocol requirements including study assessments;
* 3. Bilateral foot ulcers

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 328 (Actual)
Dates: Start 2023-04-19 (Actual); Primary Completion 2024-05-07 (Actual); Study Completion 2024-05-07 (Actual)

PRIMARY OUTCOMES:
Vibration Perception Threshold (volts) as measured by Health Care Professionals | Baseline
  Measured using Neurothesiometer and NERVE device
Vibration Perception Threshold (volts) as measured by Health Care Professionals | Follow up within baseline visit
  Measured using Neurothesiometer and NERVE device
Vibration Perception Threshold (volts) as measured by person with diabetes | Baseline
  Measured using NERVE device
Vibration Perception Threshold (volts) as measured by person with diabetes | Follow up within baseline visit
  Measured using NERVE device

CONTACTS AND LOCATIONS:
Locations (1):
- Royal Bournemouth Hospital, Bournemouth, Dorset, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided